CLINICAL TRIAL: NCT06569004
Title: Karadeniz Technical University - Tubitak Student Project
Brief Title: IR Beam Used Before Peripheral Intravenous Catheter Application on Vein Visibility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Sule BIYIK BAYRAM, Associate professor Karadeniz Technical University, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Karadeniz Tek. Univ. 3
Record Dates: First submitted 2024-01-15; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Questionnaire
Keywords: vein; intravenous; nurse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IR beam used before peripheral intravenous catheter application on vein visibility (Experimental): IR beam application
  Interventions: Device: randomised study, two group (experimental and control)
- control (No Intervention): Only parenteral catheter application

INTERVENTIONS:
Device: randomised study, two group (experimental and control) — Use of IR beam before peripheral intravenous catheter application
  Other Names: IR beam
  Arms: IR beam used before peripheral intravenous catheter application on vein visibility

SUMMARY:
The study will be conducted in the Oncology and Cardiovascular Surgery (CVS) services of a university hospital. In the research, 30 patients will constitute the control group and 30 patients will constitute the experimental group. A nurse working in the clinics where the study will be conducted will perform the PIVK procedure, and we will randomly select the control and experimental groups and apply light to the area where the PIVK will be applied to the patients in the experimental groups with a flashlight that emits infrared rays for 10 minutes. The nurse will not be aware of whether the radiation application was made to the patient or not. The veins will be evaluated by the nurse performing PIVK. We will fill out the necessary forms in ANNEX 1 (control group) and APPENDIX 2 (experimental group) while the PIVK procedure is applied. After the procedure is completed, the patient's pain, anxiety and satisfaction level during the procedure will be marked. The data will be entered into the SPSS program and evaluated with statistical tests. According to the results, the effect of IR rays used before PIVK application on the patient's pain, anxiety and satisfaction and on the procedure time spent by the nurse for the application will be determined.

DETAILED DESCRIPTION:
A nurse from the ward where the study will be conducted will be contacted and a meeting of approximately 20 minutes will be held about the study. The nurse will fill out the forms before and after inserting the catheter into the patient. Routine procedures such as tourniquet, hand opening and closing will be applied to the control group before catheter application. In the experimental group, catheter application will be made after the IR beam is applied.

ELIGIBILITY:
Inclusion Criteria:

Are between the ages of 18-70,

* PIVK will be inserted,
* Not receiving anticoagulant treatment,
* Does not have diabetes or peripheral neuropathy,
* No signs of infiltration or thrombophlebitis in the extremity where IR beam will be used,
* Dialysis patients without arteriovenous fistula,
* Does not have any communication problems and whose mental level does not cause any problems in participating in the research,
* Patients who volunteer to participate in the research will be recruited.

Exclusion Criteria:

* Sudden movements during PICK insertion,
* Missing patient data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Effect of IR beam used before peripheral intravenous catheter application | 6 mounths
  question form

SECONDARY OUTCOMES:
Effect of IR beam on pain | 6 mounths
  Pain scale
Effect of IR beam on anxiety | 6 mounths
  Anxiety scale
Effect of IR beam on satisfaction | 6 mounths
  Satisfaction scale
Effect of IR beam on application | 6 mounth
  Question form

CONTACTS AND LOCATIONS:
Overall Officials: Sule BIYIK BAYRAM, Study Director — Karadeniz Technical University
Locations (3):
- Turkey (Türkiye) (3):
  - Şule BIYIK BAYRAM, Trabzon, Ortahisar
  - Şule, Trabzon
  - Karadeniz Technical University Faculty of Health Sciences, Trabzon, Üniversite

IPD SHARING:
Plan to Share IPD: No